CLINICAL TRIAL: NCT06858137
Title: Efficacy and Safety of Thread Embedding Acupuncture for Rhinitis Allergy: Randomized Controlled Trial
Brief Title: Thread Embedding Acupuncture For Rhinitis Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2466/ĐHYD-HDDD
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Rhinitis Allergic
Keywords: Rhinitis allergic; thread embedding acupuncture; traditional medicine
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The physician responsible for administering the treatments will be aware of the group assignments but remain uninvolved in the evaluation of outcomes and subsequent data analysis. Those responsible for outcome assessment and data analysis will be kept blinded to the treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thread embedding acupuncture + fluticasone propionate spray (Experimental): Thread embedding acupuncture (TEA) every two weeks in four weeks (two sessions). Combined with fluticasone propionate spray (INCS) when needed in four weeks and lifestyle changing
  Interventions: Other: Thread embedding acupuncture; Other: Standal treatment
- fluticasone propionate spray (Active Comparator): Fluticasone propionate when needed in four weeks combined lifestyle changing
  Interventions: Other: Standal treatment

INTERVENTIONS:
Other: Thread embedding acupuncture — Thread embedding acupuncture is performed every two weeks in four weeks using a single Polydioxaone thread. Needles have a gauge size of 30G, a shaft length of 26mm, folded in half, and are applied to nine acupoints, including Yintang (EX-HN3), Yingxiang (LI20) on both sides of the body. Needles with a gauge size of 29G, a shaft length of 30mm, and a thread length of 50mm, folded in half, are used for three acupoints, which included Hegu (LI4), Zusanli (ST36), Feishu (BL13), on both sides of the body. After the thread being inserted into the body, the needle will be withdrawn immediately.
  Arms: Thread embedding acupuncture + fluticasone propionate spray
Other: Standal treatment — Inhaled corticosteroid spray - fluticasone propionate patients were permitted to use Fluticasone propionate 1 or 2 sprays (50 mcg/spray) in each nostril once a day as needed in four weeks and participants must change life style attaches including smoke and traffic pollution avoidant, preventing pets going into the bedroom, washing clothes.

SUMMARY:
Rhinitis allergy is chronic non-communicable disease with a rapid increase in the number of patients since 1990s. Rhinitis allergy is one of the risk factors for various chronic others including asthma, sinusitis, otitis media, as well as some conditions sleep disorders, emotional disorders related.

There are numerous pharmacological and non-pharmacological therapies that have been employed in management of these condition. Among them, thread embedding acupuncture (TEA) has been a widely used and established method for various chronic diseases, demonstrating its effectiveness, safety, and convenience. Several studies have shown a significant increase in treatment when combining TEA with pharmacological or other acupuncture therapies. However, there is currently no substantial data on the application of TEA for rhinitis allergy treatment.

This study is conducted to assess the efficacy and safety of combining TEA with inhaled corticosteroid (INCS) compared with ICS monotherapy in rhinitis allergy

DETAILED DESCRIPTION:
Eligible participants with rhinitis allergy, defined according to the criteria set by Allergic Rhinitis and its Impact on Asthma (ARIA) 2008, will be enrolled and subsequently randomized into two groups: the intervention group (TEA + INCS group) and the control group (INCS), with a 1:1 allocation ratio.

In both groups, the intervention duration is four weeks, with inhaled corticosteroid (INCS) - fluticasone propionate used for four weeks in required and life style changing. For the intervention group, thread embedding acupuncture (TEA) therapy will be added every two weeks, totaling two sessions during the four-week period.

Data regarding number of symptoms, BMI, Visual Analogue Scale (VAS), Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ), Relief medication score and adverse effects will be recorded immediately following randomization and weekly thereafter over the eight-week duration.

ELIGIBILITY:
Inclusion Criteria:

* Those not participating in any other clinical trial
* Those who provide written informed consent
* Those with typical symptoms of AR, rhinorrhea, sneezing, nasal obstruction, and pruritus. These symptoms should last at least one hour most day since last two week.

Exclusion Criteria:

* Pregnancy, lactation, or recent childbirth within the past 6 months.
* Those were receiving immune therapy
* Those with other allergic diseases such as bronchial asthma or allergic purpura
* Those with nasal polyposis
* Those with heterologous protein allergy
* Those with other disorders such as AIDS, vascular malformation, hypertension, hematologic, diseases, diabetes mellitus, malignant tumor, or mental disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in nasal symtoms | Assessments conducted at randomization and after each intervention week throughout the first two-week period (Week 0, Week 1, Week 2), then Week 8.
  Visual analogue scale (VAS) consists of a 100mm long line, ranging from "no troublesome at all" to "very troublesome" AR patients mark a point that best corresponds to the severity of their symptoms since a week before or current status of disease control. Participants will mark the position on the scale that corresponds to their current.

SECONDARY OUTCOMES:
Changes in quality of life | Assessments conducted at randomization and after two-week period (Week 0, Week 2, Week 6, Week 8)
  Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) has 28 questions in seven domains (activity limitation, sleep problems, nose symptoms, eye symptoms, non-nose/eye symptoms, practical problems, and emotional function). Participants will recall to their rhinitis allergy symptoms for last two weeks to respond to each question on a seven-point scale (0 = not impaired at all; 6 = severely impaired).
Changes in relief medication | Assessments conducted at randomization and after two-week period (Week 0, Week 2, Week 4, Week 6, Week 8)
  Relief medication score including the INCS dosage per day and days per week.
Proportion of intervention-related adverse effects | Up to eight weeks
  For Thread embedding acupuncture, expected AEs encompass local discomfort, post-treatment elevation in body temperature, local hematoma or subcutaneous hemorrhage, local swelling, local induration, local pain, local redness, infection, abscess, pruritus, and anaphylaxis.
  Additionally, any unexpected AEs associated with these procedures will also be documented and monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Center HCMC - Branch no.3, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juniper EF, Guyatt GH, Griffith LE, Ferrie PJ. Interpretation of rhinoconjunctivitis quality of life questionnaire data. J Allergy Clin Immunol. 1996 Oct;98(4):843-5. doi: 10.1016/s0091-6749(96)70135-5. No abstract available. PMID 8876562
- [Background] Demoly P, Bousquet PJ, Mesbah K, Bousquet J, Devillier P. Visual analogue scale in patients treated for allergic rhinitis: an observational prospective study in primary care: asthma and rhinitis. Clin Exp Allergy. 2013 Aug;43(8):881-8. doi: 10.1111/cea.12121. PMID 23889242
- [Background] Du SH, Guo W, Yang C, Chen S, Guo SN, Du S, Du ZM, Fei YT, Zhao JP. Filiform needle acupuncture for allergic rhinitis: A systematic review and meta-analysis. J Integr Med. 2022 Nov;20(6):497-513. doi: 10.1016/j.joim.2022.08.004. Epub 2022 Aug 24. PMID 36068161
- [Background] Huang JJ, Liang JQ, Xu XK, Xu YX, Chen GZ. Safety of Thread Embedding Acupuncture Therapy: A Systematic Review. Chin J Integr Med. 2021 Dec;27(12):947-955. doi: 10.1007/s11655-021-3443-1. Epub 2021 Apr 24. PMID 33893986
- [Background] Zhang J, Zhang Y, Huang X, Lan K, Hu L, Chen Y, Yu H. Different Acupuncture Therapies for Allergic Rhinitis: Overview of Systematic Reviews and Network Meta-Analysis. Evid Based Complement Alternat Med. 2020 Apr 23;2020:8363027. doi: 10.1155/2020/8363027. eCollection 2020. PMID 32382307
- [Background] Shen M, Liu J, Wang K. Effect of Traditional Chinese Medicine on Allergic Rhinitis in Children under Data Mining. Comput Math Methods Med. 2022 Jun 1;2022:7007370. doi: 10.1155/2022/7007370. eCollection 2022. PMID 35693255
- [Background] Sheng J, Jin X, Zhu J, Chen Y, Liu X. The Effectiveness of Acupoint Catgut Embedding Therapy for Abdominal Obesity: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2019 Jun 23;2019:9714313. doi: 10.1155/2019/9714313. eCollection 2019. PMID 31341504
- [Background] Ozdoganoglu T, Songu M, Inancli HM. Quality of life in allergic rhinitis. Ther Adv Respir Dis. 2012 Feb;6(1):25-39. doi: 10.1177/1753465811424425. Epub 2011 Oct 27. PMID 22032987
- [Background] Li X, Liu Y, Zhang Q, Xiang N, He M, Zhong J, Chen Q, Wang X. Effect of catgut implantation at acupoints for the treatment of allergic rhinitis: a randomized, sham-controlled trial. BMC Complement Altern Med. 2016 Nov 10;16(1):454. doi: 10.1186/s12906-016-1400-x. PMID 27829410
- [Background] Meltzer EO, Wallace D, Friedman HS, Navaratnam P, Scott EP, Nolte H. Meta-analyses of the efficacy of pharmacotherapies and sublingual allergy immunotherapy tablets for allergic rhinitis in adults and children. Rhinology. 2021 Oct 1;59(5):422-432. doi: 10.4193/Rhin21.054. PMID 34463311
- [Background] Larenas-Linnemann DES, Domthong P, Di Francesco RC, Gonzalez-Perez R, Verma M. General practitioner and patient perspectives on intranasal corticosteroids for allergic rhinitis: Treatment duration and obstacles to adherence, findings from a recent survey. World Allergy Organ J. 2024 Jun 25;17(7):100925. doi: 10.1016/j.waojou.2024.100925. eCollection 2024 Jul. PMID 39035787
- [Background] Brozek JL, Bousquet J, Baena-Cagnani CE, Bonini S, Canonica GW, Casale TB, van Wijk RG, Ohta K, Zuberbier T, Schunemann HJ; Global Allergy and Asthma European Network; Grading of Recommendations Assessment, Development and Evaluation Working Group. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines: 2010 revision. J Allergy Clin Immunol. 2010 Sep;126(3):466-76. doi: 10.1016/j.jaci.2010.06.047. PMID 20816182
- [Background] Seidman MD, Gurgel RK, Lin SY, Schwartz SR, Baroody FM, Bonner JR, Dawson DE, Dykewicz MS, Hackell JM, Han JK, Ishman SL, Krouse HJ, Malekzadeh S, Mims JW, Omole FS, Reddy WD, Wallace DV, Walsh SA, Warren BE, Wilson MN, Nnacheta LC; Guideline Otolaryngology Development Group. AAO-HNSF. Clinical practice guideline: Allergic rhinitis. Otolaryngol Head Neck Surg. 2015 Feb;152(1 Suppl):S1-43. doi: 10.1177/0194599814561600. PMID 25644617